CLINICAL TRIAL: NCT00127413
Title: Integrated Treatment for Chronic Pain and PTSD
Brief Title: Integrated Treatment for Chronic Pain and Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: D3322-R
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pain; Posttraumatic Stress Disorder
Keywords: Chronic pain; Co-morbid; Intervention; Posttraumatic Stress Disorder; Treatment
MeSH Terms: conditions — Pain; Stress Disorders, Post-Traumatic; Chronic Pain | interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitive Behavioral Therapy - Pain (Experimental): Cognitive Behavioral Therapy targeting chronic pain
  Interventions: Behavioral: Cognitive Behavioral Therapy - Pain
- Cognitive Behavioral Therapy-Integrated (Experimental): Integrated treatment for comorbid chronic pain and PTSD
  Interventions: Behavioral: Cognitive Behavioral Therapy-Integrated
- Cognitive Processing Therapy - PTSD (Experimental): Cognitive Processing Therapy for PTSD
  Interventions: Behavioral: Cognitive Processing Therapy - PTSD
- Treat as Usual (Other): Participants received care for pain and PTSD as usual from their Primary care provider
  Interventions: Behavioral: Treat as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy - Pain — Pain treatment
  Arms: Cognitive Behavioral Therapy - Pain
Behavioral: Cognitive Behavioral Therapy-Integrated — Integrated treatment
  Arms: Cognitive Behavioral Therapy-Integrated
Behavioral: Cognitive Processing Therapy - PTSD — Cognitive processing therapy
  Arms: Cognitive Processing Therapy - PTSD
Behavioral: Treat as Usual — Treatment as usual
  Arms: Treat as Usual

SUMMARY:
The purpose of this study is to examine the efficacy of an integrated treatment for Veterans with comorbid chronic pain and posttraumatic stress disorder (PTSD). It is hypothesized that Veterans who receive the integrated treatment will report more positive outcomes than individuals who are assigned to treatment as usual, pain treatment, or PTSD treatment.

DETAILED DESCRIPTION:
Chronic pain and post-traumatic stress disorder frequently co-occur and are associated with a significant level of affective distress, physical disability, and treatment resistance. However, no empirical studies have been conducted investigating the efficacy of a treatment tailored specifically for individuals with comorbid chronic pain and PTSD.

The primary objective of this study is to evaluate the efficacy of a cognitive-behavioral therapy approach for comorbid chronic pain and PTSD. A secondary objective of this study is to examine potential mechanisms of action that might mediate treatment outcome. It is hypothesized that:

1.a) Participants receiving integrated cognitive-behavioral treatment for chronic pain and PTSD will report significantly greater improvements on measures of pain, affective distress, and physical functioning from pre-treatment to post-treatment than participants in the Cognitive Behavioral Treatment for chronic pain, Cognitive Processing Therapy (CPT) for PTSD, or Treatment as Usual (TAU) conditions

1.b) All active treatments will be more effective at promoting improved outcomes than Treatment as Usual

2) Participants receiving integrated cognitive-behavioral treatment for chronic pain and PTSD will report decreased symptoms of PTSD from pre-treatment to post-treatment when compared to participants in the other conditions.

3) Participants receiving integrated cognitive-behavioral treatment for chronic pain and PTSD will report greater maintenance of change, and greater improvements on measures of Pain, Affective Distress, Physical Functioning, and PTSD at 6 months following the completion of treatment than participants in the other three conditions

4) As a secondary/exploratory hypothesis, the researchers will examine potential mechanisms of action in treatment.

It is hypothesized that changes in these potential mechanisms will mediate treatment outcome. The proposed study is a four-treatment condition by three-evaluation period (pre-treatment, post-treatment, and 6-month follow-up) repeated measures factorial design with multiple dependent measures. Participants will be 136 patients with co-morbid chronic pain and PTSD receiving care in the VA Boston Healthcare System. Participants in the active treatment conditions will complete 11 weekly outpatient therapy sessions. A clinical psychologist with specialized training in providing both PTSD and chronic pain treatment protocols will conduct therapy in an individual format, 90 minutes in duration. Participants assigned to the TAU condition will not receive treatment beyond that provided by their primary care provider and other healthcare providers. The Cognitive Behavioral Therapy-PAIN condition will follow an adaptation of a manualized treatment protocol used by Kerns and colleagues that emphasizes identifying and modifying maladaptive thoughts and behaviors related to the experience of chronic pain. Participants in the Cognitive Processing Therapy - PTSD condition will receive a manualized treatment protocol that includes several empirically supported techniques including cognitive restructuring, exposure therapy, and skills training. Participants in the Cognitive Behavioral Therapy - Integrated condition will receive an integrated treatment for comorbid pain and PTSD including components of the pain and PTSD treatments described above.

The proposed study will address the specific objectives of the National Pain Management Strategy by helping to assure that clinicians practicing in the VA healthcare system are adequately prepared to assess and manage chronic pain effectively, especially when comorbid with PTSD. Knowledge gained from the proposed study could potentially be utilized by psychologists and other healthcare providers across the VA system nationwide who are currently engaged in Cognitive Behavioral Therapy treatment programs for chronic pain and PTSD. Given that Cognitive Behavioral Therapy has been shown to be efficacious for pain and PTSD, but not for comorbid pain and PTSD, it is imperative that a new integrated treatment be evaluated that has the potential to address the unmet needs of this large population. Thus, this study will have important implications for the delivery of pain management services to veterans and others with chronic pain and PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for participation if they have chronic pain, defined as constant pain of at least six months duration with a neurologic or musculoskeletal etiology. Patients must also meet criteria for PTSD.
* Stability of pain and anxiety medications will be required for two months prior to study entry and during the active treatment and TAU phase.

Exclusion Criteria:

* Patients with life threatening or acute physical illness (e.g., cancer).
* Current alcohol or substance abuse or dependence. Veterans who have a history of alcohol or drug dependence but who have not had problematic use in the last six months will be included in the study.
* Current psychosis or suicidal ideation.
* Individuals seeking pain treatment such as surgical interventions will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Otis, BS BA PhD, Principal Investigator — VA Boston Health Care System, Jamaica Plain
Locations (1):
- VA Boston Health Care System, Jamaica Plain, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here for more information about this study: Integrated Treatment for Chronic Pain and PTSD — http://www.ptsd.va.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If it was determined during the assessment that a participant did not meet criteria for PTSD or would be excluded based on pre-determined exclusion criteria (e.g., substance use, no pain, psychosis) then the assessment was terminated and additional study related data was not collected. This was done to reduce unnecessary participant burden.
Groups:
- Cognitive Behavioral Therapy - Integrated: Integrated treatment for comorbid chronic pain and PTSD
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy - Pain | Cognitive Processing Therapy - PTSD | Cognitive Behavioral Therapy - Integrated | Treat as Usual
Started | 12 | 10 | 13 | 7
Completed | 6 | 6 | 5 | 5
Not Completed | 6 | 4 | 8 | 2
Not completed — Lost to Follow-up | 6 | 4 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Processing Therapy-PTSD: Cognitive processing therapy for PTSD
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy - Pain | Cognitive Processing Therapy-PTSD | Cognitive Behavioral Therapy-Integrated | Treat as Usual | Total
Number analyzed (Participants) | 12 | 10 | 13 | 7 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.13 (5.6) | 49.20 (5.27) | 54.18 (7.82) | 52.40 (4.67) | 52.80 (6.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 1 | 8
  Male | 11 | 7 | 10 | 6 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 5 | 3 | 3 | 2 | 13
  White | 6 | 6 | 8 | 5 | 25
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 13 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered Assessment of PTSD
Description: This 30-item structured interview is designed to assess both the 17 symptoms of PTSD and the 8 hypothesized associated features. The scale yields a dichotomous diagnosis of PTSD, and also provides a continuous score of frequency and severity for each symptom. In addition, a behaviorally anchored probe question is provided for each symptom to increase the reliability of administration. The CAPS has excellent sensitivity (.81) and specificity (.95) (Newman, Kaloupek, & Keane, 1996). For the purpose of these analyses we examined the total CAPS score. Total CAPS scores can range from 0 to 136. Higher scores represent poorer outcome with a score of greater than 50 indicating that a person meets criteria for PTSD.
Time Frame: Pretreatment (baseline), Posttreatment (3 months), and 6 month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy - Integrated: Cognitive Behavioral Therapy - Integrated treatment for pain and PTSD
Arm/Group | Cognitive Behavioral Therapy - Pain | Cognitive Processing Therapy - PTSD | Cognitive Behavioral Therapy - Integrated | Treat as Usual
Number analyzed (Participants) | 6 | 6 | 5 | 5
units on a scale
  Pretreatment | 80.67 (16.16) | 70.83 (14.13) | 77.60 (21.98) | 74.73 (15.96)
  Posttreatment | 75.5 (25.65) | 50.50 (22.06) | 62.80 (21.27) | 47.60 (32.40)
  6 month Follow-up | 79.50 (12.94) | 52.17 (32.25) | 78.40 (18.2) | 48.40 (24.04)

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Therapy - Pain | Cognitive Processing Therapy - PTSD | Cognitive Behavioral Therapy-Integrated | Treat as Usual
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/13 | 0/7

LIMITATIONS AND CAVEATS:
Failure to engage in treatment, failure to complete treatment in a timely manner due to missed treatment sessions, and difficulty with compliance with treatment session recommendations led to lower completion rates

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes